CLINICAL TRIAL: NCT05815316
Title: Fully Hybrid 18F-PSMA PET/MRI as One-stop Approach for the Diagnosis of Clinically Significant Prostate Cancer
Brief Title: 18F-PSMA PET/MRI for the Diagnosis of Clinically Significant Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: error in the registration on clincialtrials.gov. The same clinical trial has been correctly registered with the identifier NCT 06305390
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Maria Picchio, Associate Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RF-2021-12372278
Record Dates: First submitted 2023-03-21; First posted 2023-04-18 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-PSMA-1007 (Experimental): All patients undergo the same experimental procedure
  Interventions: Drug: 18F-PSMA-1007

INTERVENTIONS:
Drug: 18F-PSMA-1007 — (3S, 10S, 14S)-1-[4-[[(2S)-4-carboxy-3-[(2S)-4-carboxy-2-(6-[18F]fluoropyridin-3- amido)butanamido]butanamido]methyl]phenyl]-3- [(naphtalen-2-yl)methyl]-1,4,12-trioxo-2,5,11,13-tetraazahexadecane- 10,14,16-tricarboxilyc acid

SUMMARY:
This project aims to evaluate the role of fully hybrid PET/MRI with 18F-PSMA and multiparametric MR imaging (mpMRI) as one-stop approach for the diagnosis of clinically significant prostate cancer (csPCa).

This prospective PET/MRI clinical evaluation will ideally reduce the number of false negative findings, while at the same time, allowing also to reduce the number of unnecessary prostate biopsies in patients with low-risk, clinically indolent PCa.

The demonstration that, compared to mpMRI alone, the use of PET/MRI with 18F-PSMA has a superior diagnostic accuracy in detecting men with csPCa will strongly support the inclusion of 18F-PSMA as pre-biopsy triage test, in addition to mpMRI in daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Men at least 18 years of age referred with clinical suspicion of prostate cancer candidate for prostate biopsy
2. Feasibility to undergo all procedures listed in protocol
3. Ability to provide written informed consent

Exclusion Criteria:

1. Prior diagnosis of prostate cancer
2. Contraindication to MRI (e.g. claustrophobia, pacemaker, estimated GFR lower or equal to 50mls/min)
3. Contraindication to prostate biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
To assess the accuracy and the predictive value of fully hybrid 18F-PSMA PET/MRI for the diagnosis of csPCa | Biopsy at day 90 (+/-90)
  Diagnostic accuracy measured with sensitivity, specificity, positive and negative predicted value
To compare the proportion of csPCa missed by 18F-PSMA PET scan or mpMRI alone | Biopsy at day 90 (+/-90)
  The number of csPCa missed by PET and MR imaging when read independently
To report the change in the detection of clinically insignificant PCa when combining mpMRI and 18F-PSMA PET, and consequently the proportion of unnecessary biopsies potentially spared. | Biopsy at day 90 (+/-90)
  Only in patients with positive mpMRI and negative 18F-PSMA PET: The proportion of clinically insignificant PCa

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/16/NCT05815316/Prot_SAP_000.pdf